CLINICAL TRIAL: NCT06659250
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR OPEN, PLACEBO CONTROLLED STUDY TO ASSESS SAFETY, TOLERABILITY AND PHARMACOKINETICS OF SINGLE AND MULTIPLE ASCENDING ORAL DOSES OF PF-06414300 ADMINISTERED AS IMMEDIATE AND MODIFIED RELEASE FORMULATIONS IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn How Different Amounts and Forms of the Study Medicine Called PF-06414300 Act in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: C5651001; NCT06659250 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-10-01; First posted 2024-10-26 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Healthy Participants
Keywords: Healthy adults; First in human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-06414300 (Experimental): Participants will receive single or multiple ascending oral doses of PF-06414300
  Interventions: Drug: PF-06414300
- Placebo (Placebo Comparator): Participants will receive matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06414300 — Participants will receive oral ascending doses.
  Arms: PF-06414300
Drug: Placebo — Participants will receive matching placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn about how different amounts of study medicine called PF-06414300 acts and is changed and eliminated from the body of healthy adult participants. The amount of PF-06414300 in blood after the medicine is taken by mouth will also be measured.

The study is seeking for participants who:

* Are male or female of 18 to 65 years of age.
* Are in good health condition.
* Have body mass index of 16 to 32 kilograms per squared meters; and a total body weight of more than 50 kilograms (110 pounds).

All participants in this study will receive either PF-06414300 or placebo (dummy pill) by chance. The study will have 2 parts; in the first part of the study (Part A), each participant will receive a total of 4 doses of PF-06414300 or placebo with at least 10 to 14 days between each dose. After each dose, participants will stay in study clinic for 4 to 5 days.

In the second part of the study (Part B), each participant will receive a total of 10 doses of PF-06414300 or placebo and participants will stay in study clinic for 14 days.

An optional Japanese cohort may be done later. The planned duration of participation from screening to follow up in Part A and B of this study is up to 12 to 14 weeks and 10 to 12 weeks, respectively.

Participants will also have their blood collected by the study doctors several times.

ELIGIBILITY:
Inclusion Criteria:

* Body mass Index (BMI) of 16-32 kg/m2; and a total body weight >50 kg (110 lb).
* Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs assessments, 12-lead ECGs and laboratory tests.
* Additional criterion for participants to be enrolled in the Japanese cohort only: Participants who have 4 Japanese biologic grandparents born in Japan; body weight >45 kg (99 lb).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular (including hypertension irrespective of age), hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Recent history of abnormal bowel movements, such as diarrhea, loose stools, or constipation, within 1 week prior to first dose.
* Previous administration of an investigational product (drug or vaccine) within 30 days or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events (AE) observed after single or multiple doses | Day 1 up to Day 28 (Part A)/Day 1 up to Day 38 (Part B)
Number of Serious AE observed after single or multiple doses | Day 1 up to Day 28 (Part A)/Day 1 up to Day 38 (Part B)
Number of participants with abnormal vital sign changes following single or multiple ascending doses | Day 1 up to Day 28 (Part A)/Day 1 up to Day 38 (Part B)
Number of Participants with Electrocardiogram (ECG) Abnormalities including QT and QTcF interval following single or multiple ascending dose | Day 1 up to Day 28 (Part A)/Day 1 up to Day 38 (Part B)
Number of participants with clinically significant laboratory values | Day 1 up to Day 28 (Part A)/Day 1 up to Day 38 (Part B)

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) Part A | Day 1 up to Day 4 (Part A)
Maximum Observed Plasma Concentration (Cmax) Part A | Day 1 up to Day 4 (Part A)
Time to Reach Maximum Observed Plasma Concentration (Tmax) Part A | Day 1 up to Day 4 (Part A)
AUClast Part B | Day 1 up to Day 10 (Part B)
Cmax Part B | Day 1 up to Day 10 (Part B)
Tmax Part B | Day 1 up to Day 10 (Part B)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5651001